CLINICAL TRIAL: NCT01156025
Title: Efficacy and Safety of GV 550 in Acute Adenovirus Keratoconjunctivitis (Phase II Pilot Study, Multicentre, International, Randomised, Double-masked, Placebo-controlled, 2x40 Patients)
Brief Title: Efficacy and Safety of GV 550 in Acute Adenovirus Keratoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Medical Director, Laboratoires Théa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTGV550-PII-11/06; 2007-002455-16 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Acute Adenoviral Keratoconjunctivitis
Keywords: GV550; Acute adenoviral keratoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GV550 (Experimental): (Ganciclovir 1.5 mg/g ophtalmic gel)
  Interventions: Drug: GV550
- Placebo (Placebo Comparator): Placebo ophtalmic gel
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GV550 — Ganciclovir 1.5 mg/g, 1 drop 10 times daily at D0 and D1 and 1 drop 5 times daily from D2 to D9 + additionnal treatment (Hyabak® eye drops: 5 times daily from D10 to D30)
  Arms: GV550
Drug: placebo — 1 drop 10 times daily at D0 and D1 and 1 drop 5 times daily from D2 to D9 + additionnal treatment (Hyabak® eye drops: 5 times daily from D10 to D30)
  Arms: Placebo

SUMMARY:
The study objective is to evaluate the efficacy and the safety of GV 550 in comparison to placebo in patients with acute adenoviral keratoconjuncivitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female aged from 18 to 80 years old
* Acute adenoviral keratoconjunctivitis

Exclusion Criteria:

* Active ocular allergy
* Ocular herpès disease
* History of bacterial conjunctivitis / blepharoconjunctivitis within the last month before the inclusion visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
efficacy of GV550 | D0 to D4
  * The evolution of the inflammation
  * The virus load by quantitative PCR

SECONDARY OUTCOMES:
efficacy of GV550
  * The assessment of the patient's symptomatology evaluation
  * The score of each subjective signs
  * The score of each objective signs
  * The occurrence of focal corneal sub epithelial infiltrates (nummular stromal infiltration)
  * The occurrence of pseudo membranes
  * The virus load between D0-D10
Ocular safety
  * To compare the ocular tolerance of GV550 eye drops versus placebo eye drops with respect of the assessment of the global local tolerance assessment by the investigator and by the patient
  * To compare the ocular safety of GV550 eye drops versus placebo eye drops with respect of the assessment of the best corrected far visual acuity and ocular Adverse Event (AE) reporting at each visit
Systemic safety
  - To compare the systemic safety of GV550 eye drops versus placebo eye drops with respect of the systemic AE reporting at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Director, Clermont-Ferrand, France